CLINICAL TRIAL: NCT03435172
Title: Safety and Feasibility of Adipose Derived Regenerative Cells (ADRCs) in the Treatment of Deep Partial Thickness and Full Thickness Thermal Wounds (RELIEF)
Brief Title: Safety and Feasibility of ADRCs Treatment To Patients With Thermal Wounds
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment rate, voluntary study suspension of the study
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RELIEF
Record Dates: First submitted 2018-02-01; First posted 2018-02-15 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Thermal Burn
Keywords: Thermal Burn; Adipose Derived Regenerative Cells; Skin Graft

STUDY DESIGN:
Intervention Model Description: Subjects will have at least one deep partial or full thickness burn wound of ≥ 250 cm2 that is to be autografted with a split thickness meshed skin graft (STSG) . The Subjects will be randomized to treatment or usual care group at 2:1 ratio. Harvested tissue will be processed in the Celution® System to isolate and concentrate ADRCs. Then the subject will be followed by peripheral intravenous delivery of ADRCs within 4 hours of completion of Celution® processing.
  Up to 15 subjects will be enrolled. Each subject will contribute up to three qualified wound areas for the analysis. Randomization will be stratified to ensure that the numbers of wounds treated with STSG are balanced across the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Group (Experimental): Device-ADRCs intravenously infusion 20 million ADRCs generated by Celution device will be intraveously infused through peripheral vein. Standard care of split thickness meshed skin graft (STSG) will be used.
  Interventions: Device: Device-ADRCs intravenously infusion
- Usual Care (No Intervention): Standard care of split thickness meshed skin graft (STSG) will be used.

INTERVENTIONS:
Device: Device-ADRCs intravenously infusion — Medical Device: ADRCs Generated by Celution 800 IV Device and then Infused into Peripheral Vein.
  Arms: Treatment Group

SUMMARY:
The primary objective of the protocol is to evaluate preliminary safety and feasibility of ADRCs via intravenous delivery in the treatment of deep partial and full thickness thermal wounds.

DETAILED DESCRIPTION:
The RELIEF Trial is a prospective, open-label, parallel group, usual care controlled, multi-center randomized (2:1, active: usual care alone) safety and feasibility study targeting thermal burns. Subjects will have at least one deep partial or full thickness burn wounds of > 250 cm2 that is to be autografted with a split thickness meshed skin graft (STSG). Subjects randomized to ADRCs will undergo small volume fat harvest (100 to 150 mL) performed at initiation of general anesthesia for scheduled burn surgery followed by intravenous delivery of ADRCs within 4 hours following surgery. The lipoaspirate will be processed in the Celution® System to isolate and concentrate ADRCs.

Following informed consent and initial screening assessments, eligible subjects will undergo pre-operative testing. On the procedure day, subjects will be randomized to ADRCs (with usual care) or usual care alone. Low volume lipoharvest will only be performed on subjects randomized to ADRCs in order to obtain 100-150 mL lipoaspirate, which will then be transferred to the Celution® System for processing to isolate and concentrate ADRCs for same-day administration. All treatment will be delivered in a total volume of 10 mL which will be delivered by slow intravenous administration into a peripheral vein.

Following surgery, subjects will be evaluated at first dressing change, day 10 (±2) (only if wound dressing change planned) and weeks 2 (±3 days), 3 (±3 days), 4 (±3 days), 8 (±7 days), 12 (±14 days), 26 (±14 days), and 52(±21 days).

The 1st 5 subjects enrolled in active treatment will be observed for adverse events over a 7 day period. If no SAEs occur during that period, for that individual subject, the next subject enrolled in active treatment may be entered with the same 7 day observation period. The safety results of the first 5 subjects will be reviewed by the DMC and their evaluation will be used in conjunction with the clinical data collected to date, and if appropriate, to potentially remove the staggering approach to the study. Enrollment after the first 5 subjects may continue only after the DMC has completed its safety review and recommends continuation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age ≥ 18 to ≤ 65
* BMI > 20 kg/m2
* Burn TBSA 20% - 50%
* At least one deep partial thickness and/or full thickness thermal burn ≥ 250 cm2 on the arms, legs, back, abdomen or chest that is anticipated to be covered with autologous meshed STSG meshed and that has not been treated previously with a biologic dressing such as Alloderm® or Integra®
* Ability to safely undergo tissue harvest that is anticipated to yield >150mL of adipose tissue at a site that is free from infection
* Donor site availability for skin graft harvest
* Able to provide written informed consent signed by either the patient or their legally authorized representative
* Women and men of child-bearing potential agreeing to use contraception during the study. Acceptable methods include surgical sterility, IUDs, hormonal contraception or double barrier methods

Exclusion Criteria:

* Subjects with burns > 3rd degree (i.e. involvement of deeper tissues, such as muscle, tendons, or bone)
* Subjects with electrical or chemical burns
* Subjects with significant inhalation injuries necessitating intubation and mechanical ventilation or requiring > 50% FI02 on a continuous basis to maintain oxygenation (02 sat > 90%)
* In the opinion of treating physician, patient not expected to survive beyond 30 days
* Pre-existing condition requiring current use of immunosuppressive medication or systemic steroids
* Pregnant or lactating status. Pregnancy as determined by a positive pregnancy test at screening or baseline
* Known history of HIV infection, or active Hepatitis B or active Hepatitis C infection
* Cancer requiring chemotherapy or radiation within previous 6 months or resection within the last 5 years (other than basal cell carcinoma)
* Known chronic renal failure (serum creatinine > 2 mg/dL) or chronic liver disease
* Pre-existing medical conditions that would interfere with wound healing (i.e.diabetic patients with Hemoglobin A1c test result ≥8%, malignancy, autoimmune disease)
* Subjects with psychiatric conditions that are anticipated to result in protocol noncompliance
* Chronic illicit drug or alcohol abuse that is anticipated to interfere with patient compliance with the protocol
* Participation in another clinical trial within 60 days of the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of obtain lipo suction with > 100mL adipose tissue, Feasibility if obtain 20 million ADRC | Procedure day only
  Feasibility will be determined as 1) the ability to obtain > 100 mL adipose tissue during the liposuction surgical procedure (up to one hour for the tissue harvesting procedure), 2) obtain ≥ 20 x 106 ADRCs confirmed by cell counting (up to 4 hours after the liposuction procedure), and 3) deliver the prepared cell dose to the subject within four hours after Celution device completed the process.
Incidence of Treatment-Emergent Adverse Events [Safety] | Throughout the whole 52 weeks trial evaluation period
  Safety will be evaluated based on the incidence, type and seriousness of adverse events related to the IV administration of test substance as well as the low volume lipoharvest procedure. Adverse events will be assessed according to the NIH Common Terminology Criteria for Adverse Events (CTCAE) v4.0 for scale grading adverse events.

SECONDARY OUTCOMES:
Percent epithelialization of the graft | At first dressing change, day 10 and weeks 2, 3 and 4.
  Percent epithelialization of the graft post grafting (assessed by surgeon visual evaluation and blinded independent review of standardized photographs)
Percent take of the graft | At first dressing change, day 10 and weeks 2, 3 and 4.
  Percent take of the graft post grafting (assessed by surgeon visual evaluation and blinded independent review of standardized photographs)
Percent of wound with complete closure | At weeks 2, 3, 4, 8 and 12
  Percent of wound closure post grafting (assessed by surgeon visual evaluation and blinded independent review of standardized photographs)

CONTACTS AND LOCATIONS:
Overall Officials: Marc H Hedrick, MD, Principal Investigator — Cytori therapeutics Inc
Locations (5):
- United States (5):
  - Maricopa IHS, Phoenix, Arizona
  - Univeristy of Southern California, Los Angeles, California
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03435172/Prot_001.pdf